CLINICAL TRIAL: NCT06026566
Title: Compatible Dose Study and Effect Observation of Remimazolam Besylate Combined With Afentanil for Awake Endotracheal Intubation
Brief Title: Compatible Effect of Remimazolam Besylate Combined With Afentanil for ATI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Qiaoqiao Xu, Associate professor and deputy chief physician, Tongji Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: TongjiHospital-Anes QQ01
Record Dates: First submitted 2023-08-17; First posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-08

CONDITIONS: Remimazolam; Awake Endotracheal Intubation
Keywords: Remimazolam; Awake Endotracheal Intubation

STUDY DESIGN:
Intervention Model Description: crisscross
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Dos of R 0.1 (Experimental): The dosage of Remimazolam Besylate is 0.1 mg/kg
  Interventions: Drug: Dos of Afentanil 50; Drug: Dos of Afentanil 60; Drug: Dos of Afentanil 70; Drug: Dos of Afentanil 80; Drug: Dos of Afentanil 90; Drug: Dos of Afentanil 100
- Dos of R 0.15 (Experimental): The dosage of Remimazolam Besylate is 0.15 mg/kg
  Interventions: Drug: Dos of Afentanil 40; Drug: Dos of Afentanil 50; Drug: Dos of Afentanil 60; Drug: Dos of Afentanil 70; Drug: Dos of Afentanil 80; Drug: Dos of Afentanil 90
- Dos of R 0.2 (Experimental): The dosage of Remimazolam Besylate is 0.2 mg/kg
  Interventions: Drug: Dos of Afentanil 30; Drug: Dos of Afentanil 40; Drug: Dos of Afentanil 50; Drug: Dos of Afentanil 60; Drug: Dos of Afentanil 70; Drug: Dos of Afentanil 80
- Dos of R 0.25 (Experimental): The dosage of Remimazolam Besylate is 0.25 mg/kg
  Interventions: Drug: Dos of Afentanil 30; Drug: Dos of Afentanil 40; Drug: Dos of Afentanil 50; Drug: Dos of Afentanil 60; Drug: Dos of Afentanil 70; Drug: Dos of Afentanil 80
- Dos of R 0.3 (Experimental): The dosage of Remimazolam Besylate is 0.3 mg/kg
  Interventions: Drug: Dos of Afentanil 20; Drug: Dos of Afentanil 30; Drug: Dos of Afentanil 40; Drug: Dos of Afentanil 50; Drug: Dos of Afentanil 60; Drug: Dos of Afentanil 70
- Dos of R 0.35 (Experimental): The dosage of Remimazolam Besylate is 0.25 mg/kg
  Interventions: Drug: Dos of Afentanil 20; Drug: Dos of Afentanil 30; Drug: Dos of Afentanil 40; Drug: Dos of Afentanil 50; Drug: Dos of Afentanil 60; Drug: Dos of Afentanil 70

INTERVENTIONS:
Drug: Dos of Afentanil 20 — the dosage of Afentanil is 20 ng/ml for TCI
  Other Names: Afentanil 20
  Arms: Dos of R 0.3; Dos of R 0.35
Drug: Dos of Afentanil 30 — the dosage of Afentanil is 30 ng/ml for TCI
  Other Names: Afentanil 30
  Arms: Dos of R 0.2; Dos of R 0.25; Dos of R 0.3; Dos of R 0.35
Drug: Dos of Afentanil 40 — the dosage of Afentanil is 40 ng/ml for TCI
  Other Names: Afentanil 40
  Arms: Dos of R 0.15; Dos of R 0.2; Dos of R 0.25; Dos of R 0.3; Dos of R 0.35
Drug: Dos of Afentanil 50 — the dosage of Afentanil is 50 ng/ml for TCI
  Other Names: Afentanil 50
Drug: Dos of Afentanil 60 — the dosage of Afentanil is 60 ng/ml for TCI
  Other Names: Afentanil 60
Drug: Dos of Afentanil 70 — the dosage of Afentanil is 70 ng/ml for TCI
  Other Names: Afentanil 70
Drug: Dos of Afentanil 80 — the dosage of Afentanil is 80 ng/ml for TCI
  Other Names: Afentanil 80
  Arms: Dos of R 0.1; Dos of R 0.15; Dos of R 0.2; Dos of R 0.25
Drug: Dos of Afentanil 90 — the dosage of Afentanil is 90 ng/ml for TCI
  Other Names: Afentanil 90
  Arms: Dos of R 0.1; Dos of R 0.15
Drug: Dos of Afentanil 100 — the dosage of Afentanil is 100 ng/ml for TCI
  Other Names: Afentanil 100
  Arms: Dos of R 0.1

SUMMARY:
1. To study the pharmacokinetics between remimazolam besylate and alfentanil;
2. To determine the optimal dosage of the two drugs in awake endotracheal intubation;
3. To provide clinical guidance for awake endotracheal intubation.

DETAILED DESCRIPTION:
Tracheal intubation is the most effective and reliable method to establish artificial airway, which provides the best conditions for relieving airway obstruction, ensuring airway patency, removing respiratory secretions, preventing aspiration, assisting or controlling breathing, etc. Difficult airway management strategies must be adopted when patients are predicted to have difficulties in mask ventilation, supraglottic airway device (SAD) placement, or endotracheal intubation and front-of-neck airway (FONA) establishment. Awake tracheal intubation (ATI) is one of the important methods.

ATI refers to tracheal intubation while the patient is awake and breathing spontaneously, most commonly by flexible bronchoscopy (FB) or video laryngoscopy (VL), which allows for airway control prior to induction of general anesthesia. Thus, the potential risks and consequences of difficulty in establishing the airway after anesthesia induction are avoided. The safety of ATI is reflected in the guarantee of spontaneous breathing and intrinsic airway tension of patients before tracheal tube insertion. The failure rate of ATI is only 1-2%, and it rarely requires airway first aid or causes patient death.

ATI is currently the safest technique for dealing with difficult airways, but it accounts for only 0.2% of all tracheal intubation types in the UK. The reason is that ATI operators may be under great physical, mental, and psychological stress, which may lead to poor performance and increase the risk of complications, including failure. In addition, mechanical stimulation of the airway in the awake state can cause coughing, nausea, restlessness and other reactions to tracheal intubation, resulting in adverse consequences. Therefore, before the effective implementation of ATI, anesthesiologists often choose to combine small doses of analgesic and sedative drugs to achieve the minimum degree of sedation effect, so as to reduce the anxiety and discomfort of patients and improve the tolerance of patients.

Studies have shown that drugs such as fentanyl, remifentanil, midazolam, propofol and dexmedetomidine can be used to assist ATI to improve patient satisfaction and reduce the risk of excessive sedation and airway obstruction. However, these drugs have different degrees of cardiovascular or respiratory adverse reactions, especially when used in large doses, which increases the risk of hypoxemia, hypotension or bradycardia. ATI guidelines suggest that excessive sedation is very dangerous for some patients, and it is recommended to use it with caution, and a minimum degree of reversible sedation is preferred. Therefore, how to ensure good sedation and analgesia and maintain normal spontaneous breathing is worthy of further study.

Remimazolam besylate is a new type of benzodiazepine, which is an ultra-short-acting sedative/anesthetic drug. The mechanism is that by binding to benzodiazepine receptors, it specifically acts on GABAA receptors, enhances GABAA receptor activity, and selectively promotes extracellular chloride ions into cells, leading to hyperpolarization of cell membrane resting potential and decreased excitability, thus inhibiting neuronal electrical activity and producing sedative effect. And this effect can be specifically antagonized by flumazenil. As an important member of opioid receptor agonist, 30s of alfentanil exerts its drug effect, and its safety is far better than that of morphine. Alfentanil does not cause severe respiratory depression in the therapeutic dose range, and can reduce the use of sedative drugs when used in combination. In gastrointestinal endoscopy, hysteroscopy, fiberoptic bronchoscopy and other procedures with spontaneous breathing, alfentanil alone or in combination with benzodiazepines shows mild respiratory depression and high safety.

The purpose of this study is to study the pharmacokinetics between remimazolam besylate and alfentanil hydrochloride by response surface analysis, to determine the standard drug concentration under spontaneous breathing, and to observe the clinical effect of awake tracheal intubation under this concentration dose, to explore the best compatible dose range of the two drugs, in order to provide a reference for clinical application in patients with difficult airway.

ELIGIBILITY:
Inclusion Criteria:

1. no predictable difficult airway, Mallampati grade Ⅰ-II;
2. deviation from ideal body weight ≤25%;

   [Ideal weight (kg) = height (cm) -100 (male) or 105 (female)]
3. American Society of Anesthesiologists grade Ⅰ-II;
4. Informed consent: voluntarily participate in the trial and sign the informed consent.

Exclusion Criteria:

1. patients with head and neck lesions (including malignant tumors, previous surgery or radiotherapy), limited mouth opening, limited neck extension, obstructive sleep apnea, morbid obesity, and progressive airway injury;
2. Relative contraindications: patients with respiratory diseases, allergy to local anesthetics, airway bleeding, and non-cooperation;
3. patients known to be allergic to remimazolam besylate or benzodiazepines;
4. patients with known allergy to alfentanil or opioids;
5. body weight exceeding ±25% of ideal body weight;
6. patients with coagulation dysfunction, endocrine diseases or other hemodynamic conditions;
7. patients with a history of drug or alcohol dependence;
8. Subjects who were deemed unsuitable for the study by the investigators.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Respiratory Rate | During surgery
  RR≤8bpm means respiratory rate decreased after the use of Remimazolam Besylate and Afentanil.
Tidal volume | During surgery
  Vt≤5ml/kg means tidal volume decreased after the use of Remimazolam Besylate and Afentanil.
Deep breathing | During surgery
  Breathing hard and deep, and then PetCO2≥55mmHg mean deep breathing after the use of Remimazolam Besylate and Afentanil.
Airway obstruction | During surgery
  Difficulty in ventilation means airway obstruction after the use of Remimazolam Besylate and Afentanil.
Oxygen saturation decreased | During surgery
  SpO2≤94% means oxyfen saturation decreased after the use of Remimazolam Besylate and Afentanil.

SECONDARY OUTCOMES:
Airway status | During surgery
  Airway status evaluation during intubation
Intubation response | During surgery
  Body movement response during intubation
RASS score | During surgery
  Rass score evaluation during anesthesia induction (+4: Combative; +3: Very agitated; +2: Agitated; +1: Restless; 0: Alert and Calm; -1: Drowsy; -2: Light Sedation; -3: Moderate Sedation; -3: Moderate Sedation; -4: Deep Sedation; -5: Unarousable)
Hemodynamic assessments | During surgery
  Mean arterial blood pressure (MAP) ≤50mmHg or heart rate (HR) ≤45bpm indicates that this combination of anesthetic concentrations causes circulatory depression side effects and is recorded by "1"; otherwise, it is recorded by "0".
The satisfaction of patients and anesthesiologists | Up to 2 hours after surgery
  The satisfaction of patients and anesthesiologists with the anesthesia regimen was evaluated (very satisfied, satisfied, fair, dissatisfied, very dissatisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Qiaoqiao Xu, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong Science and Technology University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
To provide clinical application reference of the pharmacokinetics between remimazolam besylate and alfentanil for awake endotracheal intubation.
Supporting Information: Study Protocol, SAP
Time Frame: After completion of the study and publication of the article

REFERENCES:
- [Result] Bi SS, Deng CH, Zhou TY, Guan Z, Li L, Li HQ, Zhang LP, Yang L, Lu W. Remifentanil-sevoflurane interaction models of circulatory response to laryngoscopy and circulatory depression. Br J Anaesth. 2013 May;110(5):729-40. doi: 10.1093/bja/aes504. Epub 2013 Feb 6. PMID 23388507
- [Result] Ahmad I, El-Boghdadly K, Bhagrath R, Hodzovic I, McNarry AF, Mir F, O'Sullivan EP, Patel A, Stacey M, Vaughan D. Difficult Airway Society guidelines for awake tracheal intubation (ATI) in adults. Anaesthesia. 2020 Apr;75(4):509-528. doi: 10.1111/anae.14904. Epub 2019 Nov 14. PMID 31729018
- [Result] Ajay S, Singhania A, Akkara AG, Shah A, Adalja M. A study of flexible fiberoptic bronchoscopy aided tracheal intubation for patients undergoing elective surgery under general anesthesia. Indian J Otolaryngol Head Neck Surg. 2013 Apr;65(2):116-9. doi: 10.1007/s12070-012-0576-8. Epub 2012 Oct 17. PMID 24427550
- [Result] Cook TM. Strategies for the prevention of airway complications - a narrative review. Anaesthesia. 2018 Jan;73(1):93-111. doi: 10.1111/anae.14123. PMID 29210033
- [Result] El-Boghdadly K, Onwochei DN, Cuddihy J, Ahmad I. A prospective cohort study of awake fibreoptic intubation practice at a tertiary centre. Anaesthesia. 2017 Jun;72(6):694-703. doi: 10.1111/anae.13844. PMID 28654138
- [Result] Joseph TT, Gal JS, DeMaria S Jr, Lin HM, Levine AI, Hyman JB. A Retrospective Study of Success, Failure, and Time Needed to Perform Awake Intubation. Anesthesiology. 2016 Jul;125(1):105-14. doi: 10.1097/ALN.0000000000001140. PMID 27111535
- [Result] Law JA, Morris IR, Brousseau PA, de la Ronde S, Milne AD. The incidence, success rate, and complications of awake tracheal intubation in 1,554 patients over 12 years: an historical cohort study. Can J Anaesth. 2015 Jul;62(7):736-44. doi: 10.1007/s12630-015-0387-y. Epub 2015 Apr 24. PMID 25907462
- [Result] Alhomary M, Ramadan E, Curran E, Walsh SR. Videolaryngoscopy vs. fibreoptic bronchoscopy for awake tracheal intubation: a systematic review and meta-analysis. Anaesthesia. 2018 Sep;73(9):1151-1161. doi: 10.1111/anae.14299. Epub 2018 Apr 17. PMID 29687891
- [Result] Cook TM, Woodall N, Frerk C; Fourth National Audit Project. Major complications of airway management in the UK: results of the Fourth National Audit Project of the Royal College of Anaesthetists and the Difficult Airway Society. Part 1: anaesthesia. Br J Anaesth. 2011 May;106(5):617-31. doi: 10.1093/bja/aer058. Epub 2011 Mar 29. PMID 21447488
- [Result] Weinger MB, Vredenburgh AG, Schumann CM, Macario A, Williams KJ, Kalsher MJ, Smith B, Truong PC, Kim A. Quantitative description of the workload associated with airway management procedures. J Clin Anesth. 2000 Jun;12(4):273-82. doi: 10.1016/s0952-8180(00)00152-5. PMID 10960198
- [Result] Johnston KD, Rai MR. Conscious sedation for awake fibreoptic intubation: a review of the literature. Can J Anaesth. 2013 Jun;60(6):584-99. doi: 10.1007/s12630-013-9915-9. Epub 2013 Mar 20. PMID 23512191
- [Result] He XY, Cao JP, He Q, Shi XY. Dexmedetomidine for the management of awake fibreoptic intubation. Cochrane Database Syst Rev. 2014 Jan 19;2014(1):CD009798. doi: 10.1002/14651858.CD009798.pub2. PMID 24442817
- [Result] Moller IW, Krantz T, Wandall E, Kehlet H. Effect of alfentanil anaesthesia on the adrenocortical and hyperglycaemic response to abdominal surgery. Br J Anaesth. 1985 Jun;57(6):591-4. doi: 10.1093/bja/57.6.591. PMID 3924084
- [Result] Lin YJ, Wang YC, Huang HH, Huang CH, Liao MX, Lin PL. Target-controlled propofol infusion with or without bispectral index monitoring of sedation during advanced gastrointestinal endoscopy. J Gastroenterol Hepatol. 2020 Jul;35(7):1189-1195. doi: 10.1111/jgh.14943. Epub 2019 Dec 6. PMID 31802534
- [Result] Chiang MH, Wu SC, You CH, Wu KL, Chiu YC, Ma CW, Kao CW, Lin KC, Chen KH, Wang PC, Chou AK. Target-controlled infusion vs. manually controlled infusion of propofol with alfentanil for bidirectional endoscopy: a randomized controlled trial. Endoscopy. 2013 Nov;45(11):907-14. doi: 10.1055/s-0033-1344645. Epub 2013 Oct 28. PMID 24165817